CLINICAL TRIAL: NCT04679363
Title: Comparison of Active Release Technique and Post Isometric Relaxation Technique on Pain and Functional Disability in Patient With Mechanical Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/10
Record Dates: First submitted 2020-11-23; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcome assessor will be masked by withholding information related to group allocation from him
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active release technique group (Experimental): Active release technique group (ART group) will receive Oscillatory mobilization with active release technique. Treatment will be provided for 2 session/week for 3 weeks with 40 minutes/session. Patient will be assessed at baseline and after 3rd week of intervention.
  Interventions: Other: Active release technique
- Post isometric relaxation group (Experimental): Post isometric relaxation group (PIR group) will receive Oscillatory mobilization with post isometric relaxation technique. Treatment will be provided for 2 session/week for 3 weeks with 40 minutes/session. Patient will be assessed at baseline and after 3rd week of intervention.
  Interventions: Other: Post isometric relaxation

INTERVENTIONS:
Other: Active release technique — ART will be performed on upper trapezius and sternocleidomastoid, starting from 5 repetitions in 1st and 2nd week and progressing to 10 repetitions in 3rd week. ART will be performed in supine position with a pillow under knees. After the shortened area of the targeted muscle is identified, soft tissue mobilization with active movement and passive overpressure will be applied. The active movement in technique will be from shortened position of muscle to lengthened position.
  Arms: Active release technique group
Other: Post isometric relaxation — PIR will be performed on upper trapezius and sternocleidomastoid muscles, starting from 5 repetitions in 1st and 2nd week and progressing to 10 repetitions in 3rd week. The patient will be instructed to move the ear towards the shoulder of the affected side, against the resistance of the therapist's hands with minimum force (only 20% of their total force). The patient will be instructed to perform isometric contraction of the affected side along with inhalation and position for 10 seconds. Then the patient will exhale completely and relax. During this relaxation phase head and neck are taken further away from ipsilateral shoulder and ipsilateral shoulder is pushed downward until next restriction is met.
  Arms: Post isometric relaxation group

SUMMARY:
Neck pain is one of the leading causes of musculoskeletal pain and disability in the world. Despite the prevalence, accompanying disabilities, low quality of life and economic burdens of mechanical neck pain, there is a gap in high quality evidence to effectively guide the conservative treatment of this patient population. Active release technique (ART) is a soft tissue technique that focuses on removal of adhesions that build up in muscle due to overuse. ART can be used as both, as a diagnostic and treatment technique.

Limited literature is available on evaluation and treatment of neck pain by Active release technique in contrast to Post isometric release technique. This study fulfills this gap and will provide clinicians with an alternative treatment approach for mechanical neck pain.

DETAILED DESCRIPTION:
Neck pain is defined by the Global Burden of health 2010 Study as "pain in the neck with or without pain referred into one or both upper limbs that lasts for at least one day" and is one of the leading causes of musculoskeletal pain and disability in the world. Neck pain can be classified into radicular neck pain and axial neck pain. Radicular pain radiates along the nerves and is caused by irritated nerves, whereas axial pain, also called as mechanical pain, is confined to one spot or region.

Despite the prevalence, accompanying disabilities, low quality of life and economic burdens of mechanical neck pain, there is a gap in high quality evidence to effectively guide the conservative treatment of this patient population. Physical therapy management of patients with neck pain mostly include the use of treatment approaches consisting of both manual therapies including cervical spine manipulation and/or mobilization and exercise programs training for treatment of symptoms of mechanical neck pain. Active release technique (ART) is a soft tissue technique that focuses on removal of adhesions that build up in muscle due to overuse. ART can be used as both, as a diagnostic and treatment technique. Post isometric relaxation technique (PIR) is a muscle energy technique that is mostly used to relax and lengthen stiff and shortened muscles. PIR uses the muscles own energy in form of isometric contractions to relax the muscle via autogenic inhibition.

A Bacon et al (2011) conducted a study on effects of ART on tension headaches and reported that ART improved the symptoms associated with tension headaches and showed good results. A study by S Joshi et al (2018) compared the effectiveness of ART and conventional physical therapy for management of upper cross syndrome and concluded that Active release technique with conventional therapy is more effective than conventional therapy alone in the management of upper cross syndrome. Similarly, S Tak et al (2013) investigated on the effects of ART on gluteus medius for chronic pain in lower back pain and concluded that ART was effective in reducing the pain symptoms in lower back.

Limited literature is available on evaluation and treatment of neck pain by Active release technique in contrast to Post isometric release technique. This study fulfills this gap and will provide clinicians with an alternative treatment approach for mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria

* Patients with diagnosed mechanical neck pain
* Having NDI score of equal to or more than 10%
* Patients having neck pain less than 8 on NPRS

Exclusion Criteria:

* Patients having non-musculoskeletal injury
* Patients with nerve root compression
* Whiplash injuries
* History of cervical or thoracic spine surgery
* Patient on pain medication for neck pain

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating scale | 3 weeks
  The Numeric pain rating scale is a tool used for measurement of pain. The Numeric pain rating scale is a tool used for measurement of pain. It is 11-point scale from 0-10, 0 = no pain and 10 = most intense pain imaginable. Reliability for NPRS is ICC = 0.67.

SECONDARY OUTCOMES:
Algometry | 3 weeks
  Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold
Cervical Range of Motion | 3 weeks
  The cervical range of motion instrument (CROM) is a device to take objective measurements of cervical ranges. The reliability for CROM is 0.63-0.90.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No